CLINICAL TRIAL: NCT03510663
Title: A Single-center, Randomized, Double-blind (for OPC-61815 and Placebo), Placebo- and Moxifloxacin Positive-controlled, 4-Period Crossover Trial to Evaluate the Effect of Single Intravenous Administration of OPC-61815 at 16 and 32 mg on QT/QTc Interval in Healthy Male Subjects
Brief Title: Phase I Study of OPC-61815
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 263-102-00005; JapicCTI-183934 (Other: Japic)
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OPC-61815 16mg (Experimental): OPC-61815 16mg will be intravenously administered once a week.
  Interventions: Drug: OPC-61815 16mg
- OPC-61815 32mg (Experimental): OPC-61815 32mg will be intravenously administered once a week.
  Interventions: Drug: OPC-61815 32mg
- Moxifloxacin (Active Comparator): 400mg tablet will be administrated once a week.
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): Placebo will be intravenously administered once a week.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: OPC-61815 16mg — OPC-61815 16mg will be intravenously administered once a week.
  Arms: OPC-61815 16mg
Drug: OPC-61815 32mg — OPC-61815 32mg will be intravenously administered once a week.
  Arms: OPC-61815 32mg
Drug: Moxifloxacin — 400mg tablet will be administrated once a week.
  Arms: Moxifloxacin
Drug: Placebos — Placebo will be intravenously administered once a week.
  Arms: Placebo

SUMMARY:
To investigate the effects of intravenous administration of OPC-61815 at 16 and 32 mg on QT/QTc interval in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) [body weight in kg / (height in m)2] of at least 18.5 kg/m2 and less than 25.0 kg/m2 as a result of at the screening examination
* Judged by the investigator or subinvestigator to be capable of providing written informed consent prior to start of any trial-related procedures and capable of complying with the procedures for this trial

Exclusion Criteria:

* Subjects with a medical history of convulsive disorder, long QT syndrome (including family history), syncope during swimming, or any other type of syncope or cryptogenic loss of consciousness
* Subjects with a serum electrolyte abnormality (hypokalemia, hypomagnesemia, hypocalcemia, etc)
* Subjects with a family history of sudden death

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Sato, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kyusyu Region, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 (ABDC): Each subject received a single dose of each of the following 4 study treatments in Periods 1 to 4 in the assigned sequence.
  A: OPC-6181 16 mg B: OPC-61815 32 mg C: placebo D: moxifloxacin
  OPC-61815 and placebo were intravenously administered in a double-blind fashion, and a moxifloxacin 400 mg tablet was orally administered with water in an open-label fashion. A washout period of at least 6 days was set between the days of investigational medicinal product (IMP) administration in a treatment period and the next treatment period.
- Sequence 2 (DACB); Sequence 3 (BCAD); Sequence 4 (CDBA); Sequence 5 (ABCD); Sequence 6 (CADB); Sequence 7 (BDAC); Sequence 8 (DCBA): Each subject received a single dose of each of the following 4 study treatments in Periods 1 to 4 in the assigned sequence.
  A: OPC-6181 16 mg B: OPC-61815 32 mg C: placebo D: moxifloxacin
  OPC-61815 and placebo were intravenously administered in a double-blind fashion, and a moxifloxacin 400 mg tablet was orally administered with water in an open-label fashion. A washout period of at least 6 days was set between the days of IMP administration in a treatment period and the next treatment period.
Period: Overall Study
Arm/Group | Sequence 1 (ABDC) | Sequence 2 (DACB) | Sequence 3 (BCAD) | Sequence 4 (CDBA) | Sequence 5 (ABCD) | Sequence 6 (CADB) | Sequence 7 (BDAC) | Sequence 8 (DCBA)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 (ABDC) | Sequence 2 (DACB) | Sequence 3 (BCAD) | Sequence 4 (CDBA) | Sequence 5 (ABCD) | Sequence 6 (CADB) | Sequence 7 (BDAC) | Sequence 8 (DCBA) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (11.4) | 27.3 (7.4) | 30.2 (7.7) | 26.5 (9.1) | 28.3 (8.4) | 30.3 (4.4) | 27.5 (4.1) | 26.2 (6.4) | 28.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Time-matched Difference Between the OPC-61815/Moxifloxacin and Placebo Data in Change From Baseline for QTcF in 12-lead Holter Electrocardiogram (ECG)
Description: For each OPC-61815 dose, the upper limit of the confidence interval (CI) for the time-matched difference in the least squares (LS) mean for the change in QT corrected for heart rate by Fridericia's formula (QTcF) from baseline compared to the placebo data was evaluated to determine if it was lower than 10 msec at all postdose time points. Using a linear mixed effect model with baseline QTcF in each treatment period as a covariate, treatment, sequence, treatment period, time point, and interaction between treatment and time point as fixed effects, and subject as a random effect, point estimates and CIs for the time-matched difference in the LS mean for the change in QTcF from baseline compared to the placebo data were calculated.
Time Frame: Baseline, 1h, 1.5h, 2h, 3h, 4h, 6h, 12h, 24h after dosing
Population: Central tendency analysis for OPC-61815 was performed for subjects in the Pharmacodynamic Analysis Set who appropriately completed all IMP treatments and for whom predose and postdose QT data are available for all 4 treatment periods. One subject was excluded from the central tendency analysis due to lack of QT data following OPC-61815 16 mg, OPC-61815 32 mg, and placebo administration.
Measure: Least Squares Mean (Standard Error); unit: msec
Groups:
- OPC-61815 16 mg: OPC-61815 16 mg was intravenously administered once a week.
- OPC-61815 32 mg: OPC-61815 32 mg was intravenously administered once a week.
- Moxifloxacin: 400 mg tablet was orally administrated once a week.
- Placebo: Placebo was intravenously administered once a week.
Arm/Group | OPC-61815 16 mg | OPC-61815 32 mg | Moxifloxacin | Placebo
Number analyzed (Participants) | 48 | 48 | 48 | 48
msec
  1 hour postdose | 0.9 (1.1) | 0.0 (1.1) | 9.9 (1.1) | -0.9 (1.1)
  1.5 hours postdose | 2.0 (1.1) | 1.3 (1.1) | 9.5 (1.1) | -0.7 (1.1)
  2 hours postdose | 1.7 (1.1) | 0.4 (1.1) | 10.8 (1.1) | -0.4 (1.1)
  3 hours postdose | -1.2 (1.1) | -2.2 (1.1) | 10.9 (1.1) | -0.6 (1.1)
  4 hours postdose | -2.6 (1.1) | -2.2 (1.1) | 11.1 (1.1) | 1.5 (1.1)
  6 hours postdose | -11.9 (1.1) | -10.8 (1.1) | 1.9 (1.1) | -8.5 (1.1)
  12 hours postdose | -9.6 (1.1) | -9.8 (1.1) | 2.6 (1.1) | -4.7 (1.1)
  24 hours postdose | -3.6 (1.1) | -2.8 (1.1) | 4.3 (1.1) | -2.7 (1.1)
Statistical Analysis 1: Comparison: OPC-61815 16 mg vs Placebo; 1 hour postdose; Test type: Superiority; Least Squares Mean Difference = 1.8, 90% CI 2-sided [-0.4 to 4.1]
Statistical Analysis 2: Comparison: OPC-61815 16 mg vs Placebo; 1.5 hours postdose; Test type: Superiority; Least Squares Mean Difference = 2.7, 90% CI 2-sided [0.4 to 4.9]
Statistical Analysis 3: Comparison: OPC-61815 16 mg vs Placebo; 2 hours postdose; Test type: Superiority; Least Squares Mean Difference = 2.1, 90% CI 2-sided [-0.1 to 4.4]
Statistical Analysis 4: Comparison: OPC-61815 16 mg vs Placebo; 3 hours postdose; Test type: Superiority; Least Squares Mean Difference = -0.5, 90% CI 2-sided [-2.8 to 1.7]
Statistical Analysis 5: Comparison: OPC-61815 16 mg vs Placebo; 4 hours postdose; Test type: Superiority; Least Squares Mean Difference = -4.1, 90% CI 2-sided [-6.3 to -1.8]
Statistical Analysis 6: Comparison: OPC-61815 16 mg vs Placebo; 6 hours postdose; Test type: Superiority; Least Squares Mean Difference = -3.5, 90% CI 2-sided [-5.7 to -1.2]
Statistical Analysis 7: Comparison: OPC-61815 16 mg vs Placebo; 12 hours postdose; Test type: Superiority; Least Squares Mean Difference = -4.9, 90% CI 2-sided [-7.1 to -2.6]
Statistical Analysis 8: Comparison: OPC-61815 16 mg vs Placebo; 24 hours postdose; Test type: Superiority; Least Squares Mean Difference = -0.9, 90% CI 2-sided [-3.1 to 1.4]
Statistical Analysis 9: Comparison: OPC-61815 32 mg vs Placebo; 1 hour postdose; Test type: Superiority; Least Squares Mean Difference = 0.9, 90% CI 2-sided [-1.4 to 3.1]
Statistical Analysis 10: Comparison: OPC-61815 32 mg vs Placebo; 1.5 hours postdose; Test type: Superiority; Least Squares Mean Difference = 2.0, 90% CI 2-sided [-0.2 to 4.2]
Statistical Analysis 11: Comparison: OPC-61815 32 mg vs Placebo; 2 hours postdose; Test type: Superiority; Least Squares Mean Difference = 0.9, 90% CI 2-sided [-1.4 to 3.1]
Statistical Analysis 12: Comparison: OPC-61815 32 mg vs Placebo; 3 hours postdose; Test type: Superiority; Least Squares Mean Difference = -1.6, 90% CI 2-sided [-3.8 to 0.7]
Statistical Analysis 13: Comparison: OPC-61815 32 mg vs Placebo; 4 hours postdose; Test type: Superiority; Least Squares Mean Difference = -3.7, 90% CI 2-sided [-5.9 to -1.5]
Statistical Analysis 14: Comparison: OPC-61815 32 mg vs Placebo; 6 hours postdose; Test type: Superiority; Least Squares Mean Difference = -2.3, 90% CI 2-sided [-4.6 to -0.1]
Statistical Analysis 15: Comparison: OPC-61815 32 mg vs Placebo; 12 hours postdose; Test type: Superiority; Least Squares Mean Difference = -5.1, 90% CI 2-sided [-7.3 to -2.8]
Statistical Analysis 16: Comparison: OPC-61815 32 mg vs Placebo; 24 hours postdose; Test type: Superiority; Least Squares Mean Difference = -0.2, 90% CI 2-sided [-2.4 to 2.1]
Statistical Analysis 17: Comparison: Moxifloxacin vs Placebo; 1 hour postdose; Test type: Superiority; Least Squares Mean Difference = 10.8, 98% CI 2-sided [7.6 to 14.0]
Statistical Analysis 18: Comparison: Moxifloxacin vs Placebo; 1.5 hours postdose; Test type: Superiority; Least Squares Mean Difference = 10.2, 98% CI 2-sided [7.0 to 13.4]
Statistical Analysis 19: Comparison: Moxifloxacin vs Placebo; 2 hours postdose; Test type: Superiority; Least Squares Mean Difference = 11.2, 98% CI 2-sided [8.0 to 14.4]
Statistical Analysis 20: Comparison: Moxifloxacin vs Placebo; 3 hours postdose; Test type: Superiority; Least Squares Mean Difference = 11.5, 98% CI 2-sided [8.3 to 14.7]
Statistical Analysis 21: Comparison: Moxifloxacin vs Placebo; 4 hours postdose; Test type: Superiority; Least Squares Mean Difference = 9.7, 98% CI 2-sided [6.5 to 12.8]
Statistical Analysis 22: Comparison: Moxifloxacin vs Placebo; 6 hours postdose; Test type: Superiority; Least Squares Mean Difference = 10.4, 98% CI 2-sided [7.2 to 13.5]
Statistical Analysis 23: Comparison: Moxifloxacin vs Placebo; 12 hours postdose; Test type: Superiority; Least Squares Mean Difference = 7.3, 98% CI 2-sided [4.1 to 10.4]
Statistical Analysis 24: Comparison: Moxifloxacin vs Placebo; 24 hours postdose; Test type: Superiority; Least Squares Mean Difference = 7.0, 98% CI 2-sided [3.8 to 10.2]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the start of IMP administration up to an average of 31 days
Description: Safety Analysis Set included subjects who received at least 1 dose of IMP and had postdose safety data.
Arm/Group | OPC-61815 16 mg | OPC-61815 32 mg | Moxifloxacin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 3/47 | 5/47 | 1/48 | 2/47
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-61815 16 mg (N=47) | OPC-61815 32 mg (N=47) | Moxifloxacin (N=48) | Placebo (N=47)
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT03510663/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03510663/SAP_001.pdf